CLINICAL TRIAL: NCT00347997
Title: A Study to Evaluate the Safety and Effectiveness of the 217z Laser With Zyoptix for Lasik
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Decision made by B&L to cancel the study, no subjects enrolled.
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 385
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Last update posted 2011-12-08 (Estimated); Status verified 2011-12

CONDITIONS: Myopia; Astigmatism
MeSH Terms: conditions — Myopia; Astigmatism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- LASIK (Experimental): LASIK correction of myopia and myopic astigmatism
  Interventions: Device: 217z Laser

INTERVENTIONS:
Device: 217z Laser — LASIK correction of myopia and myopic astigmatism

SUMMARY:
A Study to demonstrate the safety and efficacy of wavefront laser refractive surgery treatments for myopia and astigmatism.

ELIGIBILITY:
Inclusion Criteria:

* Myopia with or without astigmatism.

Exclusion Criteria:

* Contraindications to LASIK.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Mohinder Merchea, OD, PhD, Study Director — Bausch & Lomb Incorporated